CLINICAL TRIAL: NCT06842069
Title: The Effect of Structured Education and Decision Support on Patient Outcomes for Patients Starting Dialysis Treatment in Emergency Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Zehra Aydin, AssistantProfessor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016.255.IRB3.166
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dialysis Education Program (DEP) (Active Comparator): Patients beginning urgent renal replacement treatment were placed into a Dialysis Education Program group (n=43) All patients in the DEP group were trained on the subjects included in the Dialysis Education Programme with two consequtive interview.
  Interview 1: In this 30-minute session, the aim of the training program was explained with an overview of CKD, sparing time for potential patient questions. The second training day was scheduled according to patients' agenda and their next hemodialysis session.
  Interview 2: RRT options were explained in the 30-minute training session, followed by interactive discussion with patients, ensuring that patients understood the information. When the training was completed, a guidebook ("Treatment Options in Kidney Failure-Conscious Start") was distributed to participants
  Interventions: Behavioral: Dialysis Education for Urgent Dialysis Start Patient
- Decision Tree Supported Education Program group (n=43) (Experimental): Patients beginning urgent renal replacement treatment were placed into a Decision Tree Supported Education Program group (n=43) All patients were trained on the subjects included in the Dialysis Education Programme with three consequtive interview.
  Interview 1: In this 30-minute session, the aim of the training program was explained with an overview of CKD, sparing time for potential patient questions. The second training day was scheduled according to patients' agenda and their next hemodialysis session.
  Interview 2: RRT options were explained in the 30-minute training session, followed by interactive discussion with patients, ensuring that patients understood the information. When the training was completed, a guidebook ("Treatment Options in Kidney Failure-Conscious Start") was distributed to participants Interview 3: Developed DecisionTree application ("My Life, My Choice") was performed . RRT options were assessed interactively during further discussions (30 minutes)
  Interventions: Behavioral: Decision Aid Supported Education

INTERVENTIONS:
Behavioral: Decision Aid Supported Education — Dialysis Education
  Arms: Decision Tree Supported Education Program group (n=43)
Behavioral: Dialysis Education for Urgent Dialysis Start Patient — Education provided in two consequtive educational session. During first 30-minute session, the aim of the training program was explained with an overview of CKD, sparing time for potential patient questions. The second training day was scheduled according to patients' agenda and their next hemodialysis session.
  Second Interview: RRT options were explained in the 30-minute , followed by interactive discussion with patients, ensuring that patients understood the information. When the training was completed, a guidebook ("Treatment Options in Kidney Failure-Conscious Choice, Conscious Start") was distributed to participants. The third interview date and time was scheduled with the patients in the DTSEP group.
  Arms: Dialysis Education Program (DEP)

SUMMARY:
Aim: This study aimed to develop a decision supported education program and evaluate the effect on the following dialysis patient outcomes: treatment satisfaction, treatment adherence, self-care, quality of life, depression, patient laboratory results, and clinical results.

Design: This study used a randomized controlled design. Method: Dialysis Education and Decision Tree Support application developed. Patients who started renal replacement treatment in urgent condition were placed into a Dialysis Education Program group (n=43) and Decision Tree Supported Education Program group (n=43) using the simple random sampling method. Training was provided to both groups using curriculum and training tools during two interviews. The decision tree application was used during an additional third interview with the patients in the "Decision Tree Supported Education Program" group. Data collected using the "Demographical and Clinical Data" form, the "Patient Assessment of Chronic Illness Care-Patient" Scale, the "Self-Care Ability of Chronic Dialysis Patients Assessment Scale," the "General Quality of Life Scale," and the "Patient Health Survey."

DETAILED DESCRIPTION:
Hypotheses of the study H1) A structured DTSEP improves clinical and biochemical outcomes in dialysis patients.

H2) A structured DTSEP improves treatment adherence in dialysis patients. H3) A structured DTSEP improves satisfaction in dialysis patients. H4) A structured DTSEP improves disease management in dialysis patients. H5) A structured DTSEP increases self-care competence in dialysis patients. H6) A structured DTSEP has a positive effect on patients' quality of life. H7) A structured DTSEP reduces the incidence of depression in dialysis patients.

METHOD Design and setting This experimental study used a randomized controlled design.

Participants and data collection The universe of this study consisted of patients started dialysis treatment under emergency conditions in public and private hospitals within the last one year. After predicting an effect size of 0.80 (alpha 0.05), 86 patients were included in the study. Patients were divided into a "Dialysis Education Program" (DEP) only group (n=43) and a "Decision Tree-Support Education Program" (DTSEP) group (n=43) using simple sequential sampling method. A homogenity test was performed to ensure that the patients in both groups were similar.

Inclusion criteria: Inclusion criteria required that patients: were >18 years of age, had been diagnosed with an emergent indication for dialysis treatment, displayed ESRD symptoms or signs and a glomerular filtration rate (GFR) of 5-10 mL/min/1.73 m2) (Nesrallah et al., 2014), had completed at least three hemodialysis sessions, had no problems with communication, and consented to participate in the study. Illiterate patients and those who had previously undergone RRT were excluded from the study.

Measures Socio-demographic characteristics were included in the patient information form prepared by the investigator. This form included information about patients' age, gender, marital status, education level, place of residence, economic status, and transportation to the hospital Clinical and biochemical outcomes include measurements of hemoglobin, hematocrit, albumin, total protein, C-reactive protein (CRP), calcium, phosphorus, parathormone, blood urea nitrogen (BUN), creatinine, blood pressure, residual urine volume, and Kt/V.

Treatment adherence was measured using the End Stage Renal Disease Adherence Questionnaire (ESRD-AQ), which consisted of four subgroups (adherence to total dialysis sessions, medications, fluid restrictions, and dietary recommendations), with higher scores indicating increased adherence Treatment satisfaction was measured using the Renal Treatment Satisfaction Questionnaire (RTSQ), which contained 11 questions assessing comfort, flexibility, freedom, and satisfaction with the current treatment. Higher scores in the RTSQ indicated increased satisfaction Patient Assessment of Chronic Illness Care Scale-Patient Form (Turkish PACIC): This 20-item Likert-type scale consists of five sub-dimensions: patient participation, decision-making, goal setting/guidance, problem solving, and monitoring/coordination. Higher scale score indicates that individuals with chronic disease are satisfied with the care they receive and that chronic disease management is adequate Self-Care Ability Scale for Chronic Dialysis Patients: This scale was developed by Ören in 2010 for hemodialysis and peritoneal dialysis patients . It is a triple Likert-type scale scored between 0-2 and consists of 25 items. The scores obtained from the scale range between 0-44, with drug usage scores ranging between 0-12 points, diet between 0-10, self-monitoring between 0-8, hygenic care between 0-4, and mental state between 0-6. Higher scores indicate better self-care ability of patiens

Overall Quality of Life Scale (EQ-5D):

The EQ-5D is a general health scale used to measure quality of life. The scale consists of two parts. Part A., the EQ-5D index scale, consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The index score ranges -0.59 to 1. In the score function, a value of 0 indicates death, and a value of 1 indicates perfect health. Part B. the EQ-5D VAS scale, is a visual analog scale in which individuals give values between 0 and 100 about their current health status and mark it on a thermometer-like scale. Quality of life scores range from 0-100 Patient Health Questionnaire (PHQ-9): The Patient Health Questionnaire-9 (PHQ-9) is a survey that aims to make a psychological assessment of patients in the last two weeks of dialysis, measuring the extent to which such problems disturb patients. The first part of the questionnaire consists of nine items and indicates different levels of assessment of anxiety, eating, fatigue, and somatoform changes. Each item in this section is evaluated with a 4-point Likert scale and is scored as "never" (0), "some days" (1), "more than half of the days" (2), and "almost every day" (3). A score of 1-4 points indicates minimal depression, 5-9 points indicate mild depression, 10-14 points indicate moderate depression, 15-19 points indicate moderately severe depression, and 20-27 points indicate severe depression.

Training intervention Preparation of the Dialysis Education Program A focus group interview was conducted with patients (n=14), and feedback gathered from the healthcare team (n=104) was collected by questionnaire. Preliminary results indicated that patients initiating dialysis treatment under emergency conditions lack training and decision support regarding treatment options and pre-dialysis training practices.

This analysis facilitated the preparation of the DEP (training curriculum, training booklet, training set) and development of a decision tree application. The training booklet ("Conscious Choice, Conscious Start") utilized in sessions adheres to the guidelines established by the International Patient Decision Aids Standards, encompassing topics such as kidney disease and treatment alternatives, dialysis modalities, characteristics of dialysis administration, kidney transplantation, and the experience of living with kidney disease and dialysis treatments. Subsequent to the patients undergoing DEP training, a computer-based application was created for use in DT sessions, detailing the impact of each RRT option on pertinent daily living attributes categorized under three primary headings: lifestyle, health status, and family/near surroundings. The primary objective is to offer assistance and direction throughout the decision-making process (Bekker, Winterbottom, Gavaruzzi, Finderup, & Mooney, 2023).

Application of Dialysis Education Program and Decision Tree All eligible patients who consented to participate randomly assigned in a 1:1 ratio to either the DEP or DTSEP group via an online program (www.randomization.com).

All patients in the DEP and DTSEP groups were trained on the subjects included in the education programme.

The patients in the DTSEP group had a third interview after the two consecutive training sessions.

Interview 1: After informed consent was obtained from all patients, questionnaires measuring clinical and biochemical parameters were completed before applying DEP Module 1. In this 30-minute session, the aim of the training program was explained with an overview of CKD, sparing time for potential patient questions. The second training day was scheduled according to patients' agenda and their next hemodialysis session.

Interview 2: RRT options were explained in the 30-minute Module 2 training session, followed by interactive discussion with patients, ensuring that patients understood the information. When the training was completed, a guidebook ("Treatment Options in Kidney Failure-Conscious Choice, Conscious Start") was distributed to participants. The third interview date and time was scheduled with the patients in the DTSEP group.

Interview 3: In this 30-minute session, DT application ("My Life, My Choice") was performed with patients in the DTSEP group. RRT options were assessed interactively during further discussions (30 minutes).

After completion of these sessions, all patients were scheduled to perform a third month face-to-face re-interview, using questionnaires .

Data Analysis Descriptive data were recorded using numbers and percentages or means and standard deviations, where applicable. Normality of the continuous variables were assessed by skewness and kurtosis parameters and the Kolmogorov-Smirnov test.

Homogenity of the descriptive data were evaluated using Pearson chi-square or t-test in categorical and continuous variables, respectively. Comparison of the mean differences of the two groups was performed with the t-test in independent groups if distributed normally, or the Mann Whitney U test if failed to show normal distribution.

A repeated measures analysis of variance between variables and time (pretest and posttest) in the randomized groups (DEP vs. DSDEP) was performed. A paired samples t-test was used to determine differences within groups over time. The study used an intention-to-treat analysis. This approach ensured that all randomized patients who were eligible for final testing were included in the analysis, regardless of whether they received the intervention.

Ethics Approval This study was approved by the Social Sciences Research Ethics Committee of a university (Ethics committee approval number:2016.255.IRB3.166). Institutional permissions were obtained for the study. Other permissions were acquired from the researchers who developed the questionnaire forms used in the study. Written informed consent was obtained from all patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

diagnosed with an emergent indication for dialysis treatment, displayed ESRD symptoms or signs and a glomerular filtration rate (GFR) of 5-10 mL/min/1.73 m2) completed at least three hemodialysis sessions, had no problems with communication, and consented to participate in the study.

Exclusion Criteria:

Illiterate patients and Those who had previously undergone RRT were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical and biochemical outcomes | Before intervention and one month after intervention
  Clinical and biochemical outcomes include measurements of hemoglobin, hematocrit, albumin, total protein, C-reactive protein (CRP), calcium, phosphorus, parathormone, blood urea nitrogen (BUN), creatinine, blood pressure, residual urine volume, and Kt/V
Treatment adherence | Before intervention and one month after intervention
  Treatment adherence was measured using the End Stage Renal Disease Adherence Questionnaire (ESRD-AQ), which consisted of four subgroups (adherence to total dialysis sessions, medications, fluid restrictions, and dietary recommendations), with higher scores indicating increased adherence
Patient Assessment of Chronic Illness Care Scale-Patient Form | Before intervention and one month after intervention
  Patient Assessment of Chronic Illness Care Scale-Patient Form (Turkish PACIC): Consists of five sub-dimensions: patient participation, decision-making, goal setting/guidance, problem solving, and monitoring/coordination. Higher scale score indicates that individuals with chronic disease are satisfied with the care they receive and that chronic disease management is adequate
Self-Care Ability | Before intervention and one month after intervention
  It is a data collection tool that used to asses ability of participant about medication, diet, hygenic care and mental state. Higher scores indicate better self-care ability of patiens
Quality of Life Measurement | Before intervention and one month after intervention
  The EQ-5D is a general health scale used to measure quality of life. The scale consists of two parts. Part A., the EQ-5D index scale, consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Part B. the EQ-5D VAS scale, is a visual analog scale in which individuals give values between 0 and 100
Psychological assessment | Before intervention and one month after intervention
  Aims to make a psychological assessment of patients in the last two weeks of dialysis, measuring the extent to which such problems disturb patients

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bekker HL, Winterbottom AE, Gavaruzzi T, Finderup J, Mooney A. Decision aids to assist patients and professionals in choosing the right treatment for kidney failure. Clin Kidney J. 2023 Sep 13;16(Suppl 1):i20-i38. doi: 10.1093/ckj/sfad172. eCollection 2023 Sep. PMID 37711634
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/37711634/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37711634/